CLINICAL TRIAL: NCT01669447
Title: Assessment in Early Changes in the Parameters of Optical Coherence Tomography (OCT Spectral Domain) in Patients With Subfoveal Neovascular Membranes Related to Age After Treatment With a Single Intravitreal Injection of Lucentis.
Brief Title: Evaluation of Changes in the Parameters of Optical Coherence Tomography After Intravitreal Injection of Lucentis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Osias Francisco de Souza (Other)
Responsible Party: Sponsor-Investigator, Osias Francisco de Souza, PhD in Ophthalmology, University of Campinas, Brazil
Organization: University of Campinas, Brazil (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSouza
Record Dates: First submitted 2012-08-16; First posted 2012-08-21 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Degeneration of Macula and Posterior Pole
Keywords: dmri, mnvc, lucentis
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ranibizumab (Experimental): Interventional study, prospective will be conducted in a single eye of twenty consecutive patients who will receive intravitreal ranibizumab for neovascular membrane active subfoveal choroidal active due to AMD and visual acuity of 20/40 and 20/320.
  To establish the presence of active neovascularization evaluated the presence of leakage seen on fluorescein angiography and fluid, as seen in optical coherence tomography (OCT), located both intra and subretinal, or below the retinal pigment epithelium.
  Treatment with ranibizumab will be offered after extensive Discussing the pathogenesis of AMD, the treatment alternatives, as well as the possible risks of treatment with ranibizumab. Term of consent shall be obtained prior to treatment.
  Interventions: Biological: ranibizumab

INTERVENTIONS:
Biological: ranibizumab — Interventional study, prospective will be conducted in a single eye of twenty consecutive patients who will receive intravitreal ranibizumab for neovascular membrane active subfoveal choroidal active due to AMD and visual acuity of 20/40 and 20/320.
  To establish the presence of active neovascularization evaluated the presence of leakage seen on fluorescein angiography and fluid, as seen in optical coherence tomography (OCT), located both intra and subretinal, or below the retinal pigment epithelium.
  Treatment with ranibizumab will be offered after extensive Discussing the pathogenesis of AMD, the treatment alternatives, as well as the possible risks of treatment with ranibizumab. Term of consent shall be obtained prior to treatment.
  Other Names: LUCENTIS®

SUMMARY:
Significant difference in the parameter settings of early optical coherence tomography (OCT spectal domain) in patients with subfoveal neovascular membrane realacionada age after treatment with a single intravitreal injection of Lucentis.

DETAILED DESCRIPTION:
Assessment in early changes in the parameters of optical coherence tomography (OCT spectral domain) in patients with subfoveal neovascularization secondary to age-related degeneration after treatment with a single intravitreal injection of Lucentis.

Age-related macular degeneration (AMD) leading cause of blindness over 50 years in developed Western countries. Its prevalence increases with age affecting about 8.5 to 27.9% of the population over 75 years. Its incidence has increased 30-40% in recent decades, in spite of eye diseases such as cataracts and glaucoma, which reach the same population group, have shown apparently reduced their records.

Although approximately 80% of patients with AMD have the neovascular form does not, the neovascular form is responsible for almost 90% of severe visual loss resulting from AMD. It creates great socioeconomic impact, becoming a public health problem.

Quantitative analysis of OCT has shown increasing clinical importance with the development of anti-VEGF therapy to evaluate the outcome of the treatment of neovascular AMD.

Relatively few studies in AMD has been proposed to examine the correlation between the morphological parameters of the OCT and BCVA in a systematic way.

It is important to assess the impact that different OCT parameters have on visual acuity as early as 7 days after intravitreal injection of ranibizumab in patients with AMD to define which of these parameters correlate better with the AV and prognosis. It is also unknown which patients' perception of the effectiveness of treatment in early stage. For this evaluation, we apply the visual function questionnaire (VFQ - 25) 1 and 7 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female> 50 years who signed the consent form BCAV of 20/40 20/320 (Snellen equivalent determined using ETDRS)Have choroidal neovascularization associated with AMD, have lesions involving the fovea assessed using fluorescein angiography and fundus Background of subfoveal choroidal neovascularization from the recent developments have constructive AMD disease, observed by the presence of blood, decrease the AV recent or most recent increase in the diameter range of 10% or more.

Exclusion Criteria:

* Concomitant diseases or eye conditions eye disorders that may confound interpretation of study results affecting visual acuity or require medical surgical interventions during 30 days of the study period, including retinal vascular occlusion,retinal detachment and macular hole. Eye Treatments with laser photocoagulation panretiniana eye studied for 6 months or less or focal / grid photocoagulation in the eye studied for less than 3 months of the entry into the study treatment with anti-angiogenic or intravitreal steroids in the eye studied until 4 months before randomization Any intraocular surgery on the eye studied until 3 months before History randomization vitrectomy eye conditions studied in ocular studied eye requiring concomitant therapy with corticosteroids oral or topical. Condition Treatment or systemic history of disease, metabolic dysfunction, physical examination findings, or laboratory suspected to cause disease or condition that contraindicates the use of study drugs, change the interpretation of the study or place the patient in risk of complications from the treatment. And intractable severe hypertension (diastolic blood pressure> 160 mmHg or diastolic> 100 mmHg) Use of drugs known to be toxic to the lens, retina or optic nerve including Deferoxamine, chloroquine, tamoxifen, fenotiazines, and ethambutol. Known hypersensitivity to ranibizumab or its components prior Administrative Participation of patients in studies clinical investigative drug (excluding vitamins and minerals) at 6 months (or period corresponding to five half-lives of drug investigated is greater) before randomization Failure to comply with study procedures or follow-up

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-09; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: NICOLLE ALMEIDA, GRADUATE, Study Director — CENTRO MÉDICO OFTALMOLÓGICO; Osias Souza, PI, Principal Investigator — CENTRO MEDICO OFTALMOLÓGICO; Claudia Viana, graduate, Study Chair — Centro Medico Oftalmológico
Locations (1):
- Centro Médico Oftalmológico, Campinas, São Paulo, Brazil